CLINICAL TRIAL: NCT00851864
Title: Weight-Adjusted Dosing of Tinzaparin in Pregnancy
Brief Title: Safety and Efficacy of Therapeutic Anticoagulation With Tinzaparin During Pregnancy Via Weight-based Dosing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Principal Investigator, Dr. Sue Ross, Adjunct Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 05161977
Record Dates: First submitted 2008-11-18; First posted 2009-02-26 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Venous Thromboembolism
Keywords: anticoagulation; pregnancy
MeSH Terms: conditions — Venous Thromboembolism | interventions — Tinzaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Women requiring therapeutic anticoagulation, singleton pregnancy,<30weeks
  Interventions: Drug: Tinzaparin

INTERVENTIONS:
Drug: Tinzaparin — LMWH (tinzaparin-Innohep, Leo Pharma A/S) 175 anti-factor Xa units per kilogram of body weight sub-cutaneously once daily.
  Treatment will be done for the duration of the pregnancy.
  Other Names: innohep

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of therapeutic anticoagulation with tinzaparin during pregnancy via weight-based dosing.

DETAILED DESCRIPTION:
Physicians in the Calgary Health Region are using tinzaparin (predominantly) and other low molecular weight heparins (LMWHs) for the treatment venous thromboembolism (VTE) in pregnancy. The most recent anticoagulation guidelines from American College of Chest Physicians (ACCP) suggest that heparin levels (anti-Factor-Xa activity levels) may be done periodically through pregnancy to determine the need to adjust the dose of LMWH as pregnancy progresses. This monitoring is widely practiced. There is no clear consensus in the literature, however, with some experts suggesting that initial and subsequent dosing may be done based on weight alone (as is done in the non-pregnant population). Given the multiple physiologic changes which occur to drug metabolism during pregnancy, this bears further evaluation. To date, there is very limited data on weight-adjusted dosing of LMWH in pregnancy. This study is therefore designed to determine if dosing of tinzaparin during pregnancy based on weight, with periodic weight-based adjustments, will result in adequate therapeutic anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies in women over the age of 18 requiring anticoagulation for acute VTE (DVT/PE), or high-risk prophylaxis at a tinzaparin dose of 175 IU/kg.
* High-risk patients include those with multiple (two or more) episodes of VTE and/or women receiving long-term anticoagulants (e.g. single event with known thrombophilia; APLAs and history of venous thrombosis)

Exclusion Criteria:

* Multiple gestation\
* Prosthetic valves
* Active bleeding or other contraindication to anticoagulation therapy
* Allergy to heparin, bisulfites, or fish, history of HIT (heparin induced thrombocytopenia), severe hypertension (diastolic >130)
* Severe hepatic or renal failure
* Patients over 100kg.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2007-10; Primary Completion 2010-10 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Rate of anti-Xa levels falling outside the target range of 0.4-1.2IU/mL | anti-Xa level Day 1,28, then q4 weeks

SECONDARY OUTCOMES:
mean dosage requirement in each trimester | 1 year
rate of clinical outcomes (PE/DVT) - objective testing of DVT/PE from radiology | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gibson, M.D. FRCPC, Principal Investigator — University of Calgary; Kendra Newell, M.D., Study Chair — University of Calgary; David Sam, M.D. FRCPC, Study Chair — University of Calgary
Locations (1):
- Calgary Health Region, Calgary, Alberta, Canada

REFERENCES:
- [Result] Gibson PS, Newell K, Sam DX, Mansoor A, Jiang X, Tang S, Ross S. Weight-adjusted dosing of tinzaparin in pregnancy. Thromb Res. 2013 Feb;131(2):e71-5. doi: 10.1016/j.thromres.2012.11.018. Epub 2012 Dec 13. PMID 23245654